CLINICAL TRIAL: NCT01136278
Title: Pharmacological Interaction Between Clonidine and 3,4-methylenedioxymethamphetamine (MDMA, Ecstasy)
Brief Title: Pharmacological Interaction Between Clonidine and Methylenedioxymethamphetamine (MDMA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: EK 353/09
Record Dates: First submitted 2010-05-31; First posted 2010-06-03 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Mood Disorder; Substance-Related Disorders; Amphetamine-Related Disorders
Keywords: MDMA; norepinephrine; alpha2 receptor; Ecstasy; stimulant
MeSH Terms: conditions — Mood Disorders; Substance-Related Disorders; Amphetamine-Related Disorders | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Clonidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- clonidine, MDMA, placebo (Experimental): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has 1 arm but two (actually 4) treatment conditions in the same subject.
  Interventions: Drug: 3,4-Methylenedioxymethamphetamine; Drug: Clonidine; Drug: placebo

INTERVENTIONS:
Drug: 3,4-Methylenedioxymethamphetamine — 125 mg, single dose
  Other Names: MDMA; Ecstasy
Drug: Clonidine — 150 μg per os
Drug: placebo — capsules identical to MDMA or clonidine

SUMMARY:
The purpose of this study is to determinate the effect of a pre-treatment with centrally acting alpha2-receptor agonist clonidine on the pharmacodynamics and pharmacokinetics of 3,4-methylenedioxymethamphetamine (MDMA, "Ecstasy"). The investigators hypothesize that clonidine will attenuate the subjective and cardiovascular response to MDMA.

DETAILED DESCRIPTION:
3,4-methylenedioxymethamphetamine (MDMA, "ecstasy") is widely used by young people for its euphoric effects. MDMA releases serotonin (5-HT), norepinephrine (NE), and dopamine. It is unknown which of these monoamines mainly contributes to the subjective and physiological effects of MDMA in humans. Clonidine is a centrally acting alpha2-receptor agonist and sympatholytic which attenuates the release of NE from presynaptic nerve terminals and also lowers NE plasma concentration. To determine the role of NE in the response to MDMA in humans we test the effects of a clonidine pretreatment on the pharmacodynamics and pharmacokinetics of MDMA. We use a randomized double-blind placebo-controlled cross-over design with four experimental sessions. Clonidine (150 μg) or placebo will be administered 1 h before the administration of MDMA (125 mg) or placebo to 16 healthy volunteers. Subjective and cardiovascular responses will be repeatedly assessed throughout the experiments and plasma samples are collected for pharmacokinetics. We hypothesize that clonidine will significantly attenuate predominantly the cardiovascular response to MDMA.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient understanding of the German language
* Subjects understand the procedures and the risks associated with the study
* Participants must be willing to adhere to the protocol and sign the consent form
* Participants must be willing to refrain from taking illicit psychoactive substances during the study.
* Participants must be willing to drink only alcohol-free liquids and no xanthine-containing liquids (such as coffee, black or green tea, red bull, chocolate) after midnight of the evening before the study session. Subjects must agree not to smoke tobacco for 1 h before and 4 hours after MDMA administration.
* Participants must be willing not to drive a traffic vehicle in the evening of the study day.
* Women of childbearing potential must have a negative pregnancy test at the beginning of the study and must agree to use an effective form of birth control. Pregnancy tests are repeated before each study session.
* Body mass index: 18-25 kg/m2

Exclusion Criteria:

* Chronic or acute medical condition including clinically relevant abnormality in physical exam, laboratory values, or ECG. In particular: Hypertension (>140/90 mmHg). Personal or first-grade history of seizures. Cardiac or neurological disorder.
* Current or previous psychotic or affective disorder
* Psychotic or affective disorder in first-degree relatives
* Prior illicit drug use (except THC (Tetrahydrocannabinol)-containing products) more than 5 times or any time within the previous 2 months.
* Pregnant or nursing women.
* Participation in another clinical trial (currently or within the last 30 days)
* Use of medications that are contraindicated or otherwise interfere with the effects of the study medications (monoamine oxidase inhibitors, antidepressants, sedatives etc.)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Effect of clonidine on the subjective response to MDMA | 24 h

SECONDARY OUTCOMES:
Effect of clonidine on cardiovascular effects of MDMA | 8 h
Effect of clonidine on pharmacokinetics of MDMA | 8 h
Effect of MDMA on clonidine pharmacokinetics | 8 h
Tolerability of MDMA and clonidine | 8 h
Effect of clonidine on neuroendocrine responses to MDMA | 8 h

OTHER OUTCOMES:
Genetic polymorphisms | assessed after study completion
  Effects of genetic polymorphisms on the response to MDMA

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, Principal Investigator — Department of Internal Medicine, Division of Pharmacology & Toxicology, University Hospital Basel, Switzerland
Locations (1):
- Clinical Pharmacology & Toxicology, University Hospital Basel, Basel, Basel, Switzerland

REFERENCES:
- [Derived] Vizeli P, Liechti ME. Oxytocin receptor gene variations and socio-emotional effects of MDMA: A pooled analysis of controlled studies in healthy subjects. PLoS One. 2018 Jun 18;13(6):e0199384. doi: 10.1371/journal.pone.0199384. eCollection 2018. PMID 29912955
- [Derived] Hysek CM, Liechti ME. Effects of MDMA alone and after pretreatment with reboxetine, duloxetine, clonidine, carvedilol, and doxazosin on pupillary light reflex. Psychopharmacology (Berl). 2012 Dec;224(3):363-76. doi: 10.1007/s00213-012-2761-6. Epub 2012 Jun 15. PMID 22700038